CLINICAL TRIAL: NCT04125563
Title: Influence on Cough and Airway Symptoms by Oral Capsaicin - a Phase 2, Randomised, Placebo-controlled Clinical Study in Patients With Chronic Idiopathic Cough
Brief Title: Influence on Cough and Airway Symptoms by Oral Capsaicin
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Sahlgrenska University Hospital (Other); Vinnova (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-004463-39
Record Dates: First submitted 2019-09-02; First posted 2019-10-14 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Cough
Keywords: Cough hypersensitivity syndrome; Capsaicin cough sensitivity; Cough monitor
MeSH Terms: conditions — Cough; cough hypersensitivity syndrome | interventions — oleoresins; Capsaicin

STUDY DESIGN:
Intervention Model Description: Randomised, crossover, double blind
Who Masked: Outcomes Assessor
Masking Description: Capsules, taken orally, with standardised doses of Capsicum oleoresin corresponding to 0.4 mg pure capsaicin (from chili extract) in each capsule, will be compared to matched capsules with placebo, all capsules looking the same.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo capsules (Placebo Comparator): Soft gel capsules with placebo: Sorbitol and colorant.
  Interventions: Drug: Placebos
- Active substance - oral capsaicin in soft gel capsules (Active Comparator): This is a phase 2 clinical study in humans for therapeutic use of Capsicum oleoresin - (capsaicin) in CIC. The study has a randomised, double-blind and cross-over design. During 4 weeks the participants take either active capsules (Capsicum oleoresin), or matching placebo capsules. This period follows by 2 weeks of "wash out" and then another 4 weeks with active capsules or placebo in accordance with the trial profile below.
  Interventions: Drug: Capsicum Oleoresin

INTERVENTIONS:
Drug: Capsicum Oleoresin — The soft gel capsules used in the study are easily digested in the stomach and contain standardised doses of 0,4 mg Capsicum oleoresin with the main component capsaicin (8-methyl-N-vanillyl-6-nonenamide) (from chili extract).
  Other Names: Capsaicin
  Arms: Active substance - oral capsaicin in soft gel capsules
Drug: Placebos — Soft gel capsules filled with placebo - sorbitol and colorant.
  Arms: Placebo capsules

SUMMARY:
Study objectives

To establish whether an oral intake of Capsicum oleoresin; capsaicinoids expressed as 0.4 mg capsaicin (C18H27N03; Mw: 305.4) in each capsule (from chili extract) can desensitise the cough reflex and improve unexplained coughing.

Study period

* Estimated Start date (first patient enrolled) June 2019
* Estimated End date (last patient completed follow up) June 2020
* First data available for presentation September 2020

Investigational product/comparator

The formulation is prepared from Capsicum oleoresin. Each capsule will contend a dose corresponding to 0.4 mg capsaicin. All test methods are as per the European Pharmacopoeia for Capsicum oleoresin refined and standardised.

* The formulation is developed by Research Institutes of Sweden (RISE), Sodertalje, Sweden
* Supplier of raw material for the Capsicum oleoresin product/IMP: RANSOM; Ltd, London, UK
* Producer of capsules with Capsicum oleoresin and placebo: by Catalent Pharma Solutions, St Petersburg, Florida, USA
* Packing bottles of capsules with the investigational medical product (IMP) and placebo: by Apotek Produktion & Laboratorier AB (APL), Stockholm, Sweden

Study design

Capsules, taken orally, with standardised doses of Capsicum oleoresin corresponding to 0.4 mg pure capsaicin (from chili extract) in each capsule in comparison to matched capsules with placebo (sorbitol and colorant), all capsules looking the same. Four weeks of active treatment is compared to four weeks of placebo. In between there is a wash out period of two weeks.

The time frame is 24 hours + 10 weeks. During the first 24 hours the patients carry a cough recorder (Leicester Cough Monitor - LCM) and then start with 4 weeks of active treatment or placebo. This is followed by 2 weeks of wash out and then the patients start with another 4 weeks of active treatment or placebo. After this the study ends.

Collaboration

Professor Alyn Morice MD, PhD, chief physician at Hull York Medical School, University of Hull, UK. Professor Surinder Birring MD, Senior Lecturer, specialist in respiratory medicine, Imperial College, London, UK. Associate professor Alastair Ross,PhD, Chalmers University of Technology, Gothenburg, Sweden.

Study center and number of subjects planned

All clinical trials take place at the asthma and allergy clinic, Sahlgrenska University Hospital, Gothenburg, Sweden from where 60 patients with chronic idiopathic cough (CIC) are recruited.

DETAILED DESCRIPTION:
This is a phase 2 clinical study in humans for therapeutic use of Capsicum oleoresin - (capsaicin) in chronic idiopathic cough (CIC). The study has a randomised, double-blind and cross-over design. During 4 weeks the participants take either active capsules (Capsicum oleoresin), or matching placebo capsules. This period follows by 2 weeks of "wash out" and then another 4 weeks with active capsules or placebo.

The IMP

The soft gel capsules used in the study are easily digested in the stomach and contain standardised doses of Capsicum oleoresin with the main component capsaicin (8-methyl-N-vanillyl-6-nonenamide) (from chili extract). The placebo capsules are filled with sorbitol and colorant.

Capsicum oleoresin and capsaicin is found naturally in a variety of chili fruits and the use of chili peppers in food varies greatly between different parts of the world. The maximum daily intake of capsaicin from Capsicum oleoresin in the current study could be exceeded many times in countries such as Mexico and Thailand, but it does not reach that level in most Western countries.

In concordance with the known effect of topical capsaicin for neuropathic pain, the expected effect of orally taken capsaicin is desensitisation. Capsaicin desensitise the cough-sensitive transient receptor potential vanilloids one receptors (TRPV1) and other TRP receptors followed by decreased cough reflex sensitivity and coughing in patients with CIC. Capsaicin causes depletion of neuropeptides leading to "exhausting" of the receptor with ameliorated symptoms in the patients.

In the application to the Swedish Medical Products Agency the capsules, the active product ingredient (API) and the formulation are extensively described in the investigational medical product dossier (IMPD).

In summary

* Supplier of raw material for the Capsicum oleoresin product/IMP: RANSOM; Ltd, London, UK
* The IMP is developed by RISE, Sodertalje, Sweden
* Filling of capsules with Capsicum oleoresin and placebo: Catalent Pharma Solutions, St Petersburg, Florida, USA
* Packing in bottles of capsules with IMP and placebo: by Apotek Produktion & Laboratorier AB (APL), Stockholm, Sweden
* Labelling: Tamro, Gothenburg, Sweden (an independent pharmaceuticals logistics service provider). Each package will be labelled with study code, randomisation number, dosage form, quantity, dosage instructions, name of investigator, expiry date, storage instruction.
* Storage: in room temperature at the allergy clinic at Sahlgrenska University Hospital and at Tamro, Gothenburg, Sweden
* Independent monitoring of the clinical study by qualified staff from Gothia Forum, Sahlgrenska University Hospital, Gothenburg, Sweden
* A safety report will be completed after the study end and sent to the relevant Competent Authority and the Ethics Committee

Study population

60 patients with CIC from the outpatient clinic at the asthma and allergy clinic, Sahlgrenska University Hospital, Gothenburg, Sweden are included.

Study design

The total study time for each patient is 24 hours + 10 weeks and includes 6 visits. At the first visit tests and questionnaires are assessed as described below (outcome measures) and the patients collect a cough monitor to record cough during 24 hours. After returning the cough monitor the patients start with 4 weeks of active treatment or placebo. This is followed by 2 weeks of wash out and then the patients start with another 4 weeks of active treatment or placebo. After this the study ends. Estimated time for each visit is 2 hours.

During the first 2 weeks of each arm (active or placebo) of 4 weeks the patients take one capsule morning and evening. During the following 2 weeks they take 2 capsules morning and evening.

At each visit:

* The patients answer the questionnaires LCQ-S, the HARQ-S and also score their cough severity during the past two weeks using a VAS-scale (0-100 mm)
* A cough sensitivity test is performed with a standardised capsaicin inhalation test, assessing concentration of inhaled capsaicin causing 2 coughs (C2), 5 coughs (C5) and 10 coughs (C10)
* Lung function measured with spirometry and impulse oscillometry (IOS)
* Pain sensitivity is assessed with pressure algometry at 4 pre-defined points
* Levels of capsaicin/dihydrocapsaicin in sera are measured

At 4 opportunities:

1: 24 hours before any treatment. 2: at the end of 4 weeks of active treatment or placebo respectively. 3: at the end of 2 weeks wash out. 4: at the end of 4 weeks of active treatment or placebo respectively:

* Fraction of exhaled nitric oxide (FeNO) is measured
* Particles in exhaled air (PExA) are measured
* The cough frequency during 24h is assessed using the LCM cough monitor

Statistical Analysis Plan (SAP):

All detailed statistical analyses will be specified in a separate study SAP that is developed and finalized.

Sample size calculation

The sample size calculations for the primary variables LogC2 and LogC5 given the results obtained in an earlier pilot study are described in the following:

In order to reach the power of 0.80 with mean difference in LogC2 between the Active-Placebo treatment of 0.590 and standard deviation for the difference of 0.885, with two-tailed Fisher's non-parametric permutation test, alpha = 0.025, 24 patients are needed to be included in the study.

In order to reach the power of 0.80 with mean difference between in LogC5 the Active-Placebo treatment of 0.425 and standard deviation for mean difference of 0.911, with two-tailed Fisher's non-parametric permutation test, alpha = 0.025, 47 patients are needed to be included in the study.

In order to adjust for drop-outs, 60 patients will be included in this study. Statistical methodology The main analyses will be on the ITT population and complementary analyses will be performed on the PP population. In this cross over study all main analysis will be adjusted for period effects.

For non-normal continuous variables, ordered categorical variables and dichotomous variables the following non-parametric analyses of cross-over design for test between Capsaicin and Placebo will be used, adjusting for period effects. The difference between period 2 and period 1 values will be calculated and this difference will be tested between the treatment sequences. For continuous variables this difference will be continuous and analysed with Fisher's non-parametric permutation test. For ordered categorical variables and dichotomous variables this difference will be an ordered categorical variable and analysed with Mantel-Haenszel chi-square test.

The test regarding the effect of Capsaicin vs Placebo on normally distributed efficacy variables will be performed by using generalised linear models for cross-over design, with sequence, period and treatment group as fixed effects. SAS code for the analysis of normally distributed data:

PROC MIXED; CLASS SEQ PATIENT PERIOD TRT; MODEL Y=SEQ PERIOD TRT; REPEATED / TYPE=CS SUB=PATIENT(SEQ); RUN; The most appropriate variance-covariance structure will be used, that might by other than Compound Symmetry (CS) specified in the code above.

For continuous variables the distribution of the variables will be given at baseline, visit 2 and visit 4 and change from baseline to visit 2 and 4 by Capsaicin treatment and placebo.

95% confidence interval for the mean difference between Capsaicin and placebo treatment adjusted for period effect will be given. The results will be presented in both tables and figures.

All categorical variables will be described by number and percentage, and all continuous variables by mean, standard deviation, median, minimum and maximum.

The carry-over effect for the primary variables will be analysed by testing the mean of period 1 and period 2 values between the two treatment sequences.

For test of change within groups Sign test will be used for ordered categorical variables and dichotomous variables and Fisher's non-parametric permutation test for paired observations for continuous variables.

The missing values will be imputed by using stochastic imputation (seed=99786) using all available baseline and relevant follow-up data for all efficacy analyses.

The main analyses will be performed on stochastic imputed values and sensitivity analyses on complete case and on last observation carried forward for primary efficacy variable. Baseline and demographic variables will be described for the total sample.

The study will be considered positive in case any of the two primary variables reach the significance level below 0.025. For all other tests the significance level of 0.05 will be applied. All significance tests will be two-tailed and all analyses will be performed by using SAS® v9.4 or later (SAS Institute Inc., Cary, NC, USA).

ELIGIBILITY:
Inclusion Criteria:

* Out-patients, men and women
* Age 18-75 years
* Present non-smoker
* A diagnosis of CIC, set by a trained specialised physician
* Exceeding the cut off limit for the Swedish version of the Hull Airway Reflux Questionnaire (HARQ-S): (a total score of ≥13 points)
* At screening visit reporting daily, troublesome coughing and an easily evoked cough reflex since at least two months
* At screening visit having a positive capsaicin inhalation cough test

Exclusion Criteria:

* Known or suspected chili allergy
* Known or suspected allergy to the colorant Tartrazine (FD&C Yellow #6)
* Any kind of diabetes
* Treatment the preceding month with any kind of chili medication or food supplement containing capsaicin or having a diet including chili in treatment purpose
* Treatment the preceding month with medication according to the study protocol
* Pregnancy, breast-feeding, planned pregnancy during the study and fertile women not using acceptable contraceptive measures, as judged by the investigator
* Suspected poor capability to follow instructions of the study, e.g. because of a history of drug abuse, difficult to read and/or understand Swedish or any other reason, as judged by the investigator
* Airway infection the last 4 weeks before study start
* Any significant disease or disorder which, in the opinion of the investigator, may either put the patient at risk because of participation in the study, or influence the results of the study, or the patient's ability to participate in the study
* Any clinically relevant abnormal findings in physical examination, vital signs at baseline visit, which, in the opinion of the investigator, may put the patient at risk because of his/her participation in the study
* Previous randomisation of treatment in the present study
* Participation in another clinical study 30 days prior to and during this study
* Smoking during the last ten years or/and >10 pack years
* Known alcohol and/or drug abuse
* The participants will be asked for any season allergy or other allergy and for allergen exposure. The study start date will be adjusted to season or another possible allergen exposure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Capsaicin cough sensitivity | From baseline up to 4 weeks post-treatment.
  The primary efficacy variables will be capsaicin inhalation cough sensitivity at each visit in terms of:
  * LogC2 (logarithmic values of the inhaled capsaicin threshold concentration needed to reach two coughs (C2)). Change from baseline at the end of two and four weeks of treatment with active substance or placebo
  * LogC5 (logarithmic values of the inhaled capsaicin threshold concentration needed to reach five coughs (C5)). Change from baseline at the end of two and four weeks of treatment with active substance or placebo

SECONDARY OUTCOMES:
Cough monitor recordings | From baseline up to 4 weeks post-treatment.
  Objectively measured cough counting (LCM) at four opportunities. Change from baseline at the end of four weeks of treatment with active substance or placebo.
Visual analogue scale (VAS-scale) | From baseline up to 4 weeks post-treatment.
  At each visit: Using the VAS-scale evaluating 6 symptoms; cough, rhinitis, throat irritation, dyspnoea, stomach problems and urinary incontinence are recorded on a VAS-scale of 0 to 100 mm, with 0 indicating no symptoms and 100 indicating intense symptoms. The patients put an X on a line of exactly 100 millimeters. The nurse then measures the length from the beginning of the line to the X and register this in the case report form. There are no subscores. The patients are told that an X on the line's beginning indicates no symptoms at all and an X at the line's ending indicates worse possible symptoms.
  Change from baseline to each of the four weeks of treatment with active substance and placebo. The procedure takes about 5 minutes. The analyses for all patients will be performed when the entire study is completed.

OTHER OUTCOMES:
Height | From baseline up to 4 weeks post-treatment.
  At study start the patient's height is recorded in meters.
Weight | From baseline up to 4 weeks post-treatment.
  At each visit the patient's weight in kilograms will be recorded.
BMI - Body Mass Index. Weight and height will be combined to report BMI in kg/m2. | From baseline up to 4 weeks post-treatment.
  At each visit the patient's weight in kilograms will be recorded and aggregated with the height measured at baseline to calculate BMI in kg/m2.
Lung function: Forced expiratory volume (liters) in one second (FEV1). | From baseline up to 4 weeks post-treatment.
  At each visit the FEV1 is measured (and predicted values of FEV1 according to gender, age and body length) using the Masterscope spirometer (Masterscope, APS version 5.02 software). After a maximal inhalation a forced exhalation during one second is recorded.
Lung function: Predicted value (%) of Forced expiratory volume (liters) in one second (FEV1). | From baseline up to 4 weeks post-treatment.
  At each visit the predicted values of FEV1 according to gender, age and body length) will be calculated using the Masterscope spirometer (Masterscope, APS version 5.02 software). After a maximal inhalation a forced exhalation during one second is recorded.
Lung function: Forced vital capacity (FVC) (liters). | From baseline up to 4 weeks post-treatment.
  At each visit the FVC is measured using the Masterscope spirometer (Masterscope, APS version 5.02 software). The FVC is calculated after maximal inhalation followed by a forced maximal exhalation.
Lung function: FEV% | From baseline up to 4 weeks post-treatment.
  At each visit FEV% is measured. FEV% is defined as FEV1/VC and is thus a measure of how much of her/his vital capacity the patient exhales during the first second of a forced expiration.
Lung function: Impulse oscillometry (IOS) (Resistance - Hz) | From baseline up to 4 weeks post-treatment.
  At each visit after the spirometry is assessed lung function is also measured with impulse oscillometry (IOS) to record airway resistance at 5 and 20 hertz and to measure the area under the curve (Ax) mirroring the resistance in the peripheral airways using Jaeger Masterscope IOS™. After this the participants inhale bronchodilator medication and 15 minutes thereafter perform an additional lung function test. This is a standard procedure for examining lung function.
Lung function: Fractional exhaled nitric oxide (FeNO) | From baseline up to 4 weeks post-treatment.
  At 4 visits lung function is also evaluated with measurements of fractional exhaled nitric oxide (FeNO) in accordance with international American Thoracic Society/ERS recommendations, using a NIOX, nitric oxide gas analyser (Aerocrine AB, Stockholm, Sweden).
Cough sensitivity to inhaled capsaicin - to reach 10 coughs | From baseline up to 4 weeks post-treatment.
  At each visit: LogC10 (logarithmic values of the inhaled capsaicin threshold concentration needed to reach 10 coughs) (C10)). Change from baseline at the end of two and four weeks of treatment with active substance or placebo.
Examination of the amount, weight and composition of particles in exhaled air by the PExA method. | From baseline up to 4 weeks post-treatment.
  At each visit: Evaluating possible chemical changes in the small airways by collecting particles in the exhaled air with a non-invasive method using the PExA 2.0 (PExA AB, Gothenburg, Sweden). After capsaicin provocation and lung function measurements exhaled particles are measured with White FHLC Membrane Filter Type: 0.45mm and then frozen for later analyses.
The Swedish version of the Hull Airway Reflux Questionnaire (HARQ-S) | From baseline up to 4 weeks post-treatment.
  At each visit: The Hull Airway Reflux Questionnaire (HARQ) was developed with the aim of eliciting the major component of chronic cough in adults. It comprises 14 items with a maximum total score of 70. A Swedish version (HARQ-S) has previously been validated. A total score of <13 points is regarded as normal while higher scores indicate more symptoms and problems of chronic cough.
The Swedish version of the Leicester Cough Questionnaire (LCQ-S) | From baseline up to 4 weeks post-treatment.
  At each visit: The validated LCQ-S is a self-reporting quality of life measure of chronic cough for adults. It consists of 19 items with a 7-point response scale (range from 1 to 7). Each item is developed to assess symptoms during cough and impact of cough on three main domains: physical, psychological and social. Scores are calculated as a mean of each domain and total score is calculated by adding every domain score.
Pain sensitivity with pressure algometry (PPT) | From baseline up to 4 weeks post-treatment.
  At each visit: Pain sensitivity is evaluated by pressure pain thresholds for measuring and quantifying deep tenderness in muscles. The Somedic algometer (SBMEDIC Electronics, Solna, Sweden) is a gun-shaped handle creating pressure through a pressure sensitive strain gauge at the tip, connected to a power supply, an amplifier and a display unit. The display shows the actual pressure given (kPa/s), and a scale indicates the rate of pressure to help the examiner to keep the pressure constant.
Chest mobility | From baseline up to 4 weeks post-treatment.
  At each visit: Chest mobility (in cm) is assessed with a tape measure as chest expansion, thoracic flexion and extension. Chest expansion is measured as the circumference difference after maximal inhalation through the nose and maximal exhalation through the mouth at the level of the xiphoid process with participants in a standing position with their hands on their head. Thoracic flexion and thoracic extension are measured 30 cm distally from the seventh cervical vertebrae (C7) in a standing position with the patient's hands along their sides. Every measurement is performed three times, and the best of the three measurements is noted.
Serum analyses of capsaicin and dihydrocapsaicin | From baseline up to 4 weeks post-treatment.
  At each visits samples are taken for serum analyses with high performance liquid chromatography (HPLC) in accordance with Hartley et al:
  "Total capsaicinoids are extracted from 1 mL aliquots of serum or plasma using methyl-isobutyl ketone, evaporation of the extract to dryness and reconstitution with 200 microliter of acetonitrile. The HPLC mobile phase is 40:60 water:acetonitrile. The absorbance of the eluent is monitored at 205 nm. Inter batch reproducibility for both is 15%. The limits of detection are 2.6 and 3.8 ng/mL for capsaicin and dihydrocapsaicin respectively." Also see reference.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Millqvist, MD, PhD, Principal Investigator — Vastra Gotaland Region
Locations (1):
- Allergy clinic, Sahlgrenska University Hospital, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ternesten-Hasseus E, Johansson EL, Millqvist E. Cough reduction using capsaicin. Respir Med. 2015 Jan;109(1):27-37. doi: 10.1016/j.rmed.2014.11.001. Epub 2014 Nov 12. PMID 25468411
- [Background] Pullerits T, Ternesten-Hasseus E, Johansson EL, Millqvist E. Capsaicin cough threshold test in diagnostics. Respir Med. 2014 Sep;108(9):1371-6. doi: 10.1016/j.rmed.2014.07.012. Epub 2014 Aug 4. PMID 25129869
- [Background] Hartley T, Stevens B, Ahuja KD, Ball MJ. Development and experimental application of an HPLC procedure for the determination of capsaicin and dihydrocapsaicin in serum samples from human subjects. Indian J Clin Biochem. 2013 Oct;28(4):329-35. doi: 10.1007/s12291-013-0297-0. Epub 2013 Jan 20. PMID 24426233
- [Background] Johansson EL, Ternesten-Hasseus E, Olsen MF, Millqvist E. Respiratory movement and pain thresholds in airway environmental sensitivity, asthma and COPD. Respir Med. 2012 Jul;106(7):1006-13. doi: 10.1016/j.rmed.2012.03.011. Epub 2012 Apr 15. PMID 22510540
- [Background] Sonnerfors P, Faager G, Einarsson U. Translation of the Leicester Cough Questionnaire into Swedish, and validity and reliability in chronic obstructive pulmonary disease. Disabil Rehabil. 2018 Nov;40(22):2662-2670. doi: 10.1080/09638288.2017.1353648. Epub 2017 Jul 20. PMID 28728439
- [Background] Johansson EL, Ternesten-Hasseus E. Reliability and Validity of the Swedish Version of the Hull Airway Reflux Questionnaire (HARQ-S). Lung. 2016 Dec;194(6):997-1005. doi: 10.1007/s00408-016-9937-5. Epub 2016 Sep 16. PMID 27638152